CLINICAL TRIAL: NCT04523129
Title: A Phase 3, Multi-center, Randomized, Double-masked, Vehicle-controlled Clinical Trial to Assess the Efficacy and Safety of Topical CyclASol® for the Treatment of Dry Eye Disease
Brief Title: ESSENCE 2: CyclASol for the Treatment of Signs and Symptoms of Dry Eye Disease (DED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novaliq GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CYS-004
Record Dates: First submitted 2020-08-19; First posted 2020-08-21 (Actual); Results first posted 2023-03-10 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Ophthalmic Solutions; Cyclosporins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CyclASol Ophthalmic Solution (Experimental): Cyclosporine A solution in vehicle
  Interventions: Drug: CyclASol topical ocular, eye drops
- Vehicle Ophthalmic solution (Placebo Comparator): Vehicle only
  Interventions: Drug: Vehicle topical ocular, eye drops

INTERVENTIONS:
Drug: CyclASol topical ocular, eye drops — Cyclosporine A solution in vehicle
  Other Names: Ciclosporine (CSA)
  Arms: CyclASol Ophthalmic Solution
Drug: Vehicle topical ocular, eye drops — Vehicle
  Other Names: Vehicle
  Arms: Vehicle Ophthalmic solution

SUMMARY:
The objective of this pivotal trial is to assess the efficacy, safety and tolerability of CyclASol in comparison to the vehicle for the treatment of signs and symptoms of Dry Eye Disease (DED).

DETAILED DESCRIPTION:
This Phase 3 study will assess the efficacy, safety and tolerability of CyclASol 0.1% Ophthalmic Solution administered bilaterally twice daily versus vehicle.

ELIGIBILITY:
Inclusion Criteria:

* Signed ICF (Informed Consent Form)
* Patient-reported history of DED in both eyes
* Current use of OTC (over-the-counter) and/or artificial tears for dry eye symptoms
* Ability and willingness to follow instructions, including participation in all study assessments and visits

Exclusion Criteria:

* Women who are pregnant, nursing or planning a pregnancy
* Unwillingness to submit a urine pregnancy test at screening and the last visit (or early termination visit) if of childbearing potential, or unwillingness to use acceptable means of birth control
* Clinically significant slit-lamp findings or abnormal lid anatomy at screening
* Ocular/periocular malignancy
* History of herpetic keratitis
* Active ocular allergies or ocular allergies that may become active during the study period
* Ongoing ocular or systemic infection at screening or baseline
* Wear of contact lenses within 3 months prior to screening or anticipated use of contact lenses during the study
* Use of topical Cyclosporine A or Liftigrast within 2 months prior to screening
* Intraocular surgery or ocular laser surgery within the previous 6 months, or have any planned ocular and/or lid surgeries over the study period
* Presence of uncontrolled systemic diseases
* Presence of known allergy and/or sensitivity to the study drug or its components
* Randomized in a previous CyclASol trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 834 (Actual)
Dates: Start 2020-12-05 (Actual); Primary Completion 2021-09-03 (Actual); Study Completion 2021-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sonja Kroesser, PhD, Study Director — Novaliq GmbH
Locations (27):
- United States (27):
  - CYS-004 Investigational Site, Phoenix, Arizona
  - CYS-004 Investigational Site, Los Angeles, California
  - CYS-004 Investigational Site, Newport Beach, California
  - CYS-004 Investigational Site, Santa Ana, California
  - CYS-004 Investigational Site, Colorado Springs, Colorado
  - CYS-004 Investigational Site, Fort Lauderdale, Florida
  - CYS-004 Investigational Site, Chicago, Illinois
  - CYS-004 Investigational Site, Carmel, Indiana
  - CYS-004 Investigational Site, Indianapolis, Indiana
  - CYS-004 Investigational site, Louisville, Kentucky
  - CYS-004 Investigational Site, Andover, Massachusetts
  - CYS-004 Investigational Site, Raynham, Massachusetts
  - CYS-004 Investigational Site, Medina, Minnesota
  - CYS-004 Investigational Site, Kansas City, Missouri
  - CYS-004 Investigation Site, Kansas City, Missouri
  - CYS-004 Investigational Site, Henderson, Nevada
  - CYS-004 Investigational Site, Raleigh, North Carolina
  - CYS-004 Investigational Site, Shelby, North Carolina
  - CYS-004 Investigational Site, Fargo, North Dakota
  - CYS-004 Investigational Site, Cranberry Township, Pennsylvania
  - CYS-004 Investigational Site, Warwick, Rhode Island
  - CYS-004 Investigational Site, Memphis, Tennessee
  - CYS-004 Investigational Site, Smyrna, Tennessee
  - CYS-004 Investigational Site, Layton, Utah
  - CYS-004 Investigational site, Ogden, Utah
  - CYS-004 Investigational Site, Lynchburg, Virginia
  - CYS-004 Investigational Site, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Akpek EK, Wirta DL, Downing JE, Tauber J, Sheppard JD, Ciolino JB, Meides AS, Krosser S. Efficacy and Safety of a Water-Free Topical Cyclosporine, 0.1%, Solution for the Treatment of Moderate to Severe Dry Eye Disease: The ESSENCE-2 Randomized Clinical Trial. JAMA Ophthalmol. 2023 May 1;141(5):459-466. doi: 10.1001/jamaophthalmol.2023.0709. PMID 37022717

RESULTS

PARTICIPANT FLOW:
Groups:
- CyclASol Ophthalmic Solution: Cyclosporine A solution in vehicle
  CyclASol topical ocular, eye drops: Cyclosporine A solution in vehicle (one drop per eye BID)
- Vehicle Ophthalmic Solution: Vehicle only
  Vehicle topical ocular, eye drops: Vehicle (one drop per eye BID)
Period: Overall Study
Arm/Group | CyclASol Ophthalmic Solution | Vehicle Ophthalmic Solution
Started | 423 | 411
Completed | 415 | 402
Not Completed | 8 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CyclASol Ophthalmic Solution | Vehicle Ophthalmic Solution | Total
Number analyzed (Participants) | 423 | 411 | 834
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (15.36) | 56.6 (16.30) | 57.1 (15.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 306 | 303 | 609
  Male | 117 | 108 | 225
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 62 | 60 | 122
  Not Hispanic or Latino | 359 | 348 | 707
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 423 | 411 | 834

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Corneal Fluorescein Staining
Description: Total Corneal Fluorescein Staining (tCFS) is graded based on the National Eye Institute (NEI) scale. The NEI scale divides the cornea in 5 subregions: central, inferior, superior, nasal, temporal. The score for each region ranges from 0-3; 0 corresponds to no staining (best), 3 corresponds to maximum staining (worst). The total score is the sum of the 5 subregions ranging from 0 (best) - 15 (worst).
Time Frame: baseline and 1 month [day 29]
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | CyclASol Ophthalmic Solution | Vehicle Ophthalmic Solution
Number analyzed (Participants) | 409 | 395
score on a scale | -3.96 (0.146) | -3.55 (0.149)

2. Primary Outcome: Change From Baseline in Eye Dryness Score
Description: Eye dryness score is rated on a visual analogue scale (VAS) ranging from 0-100; 0 corresponds to no discomfort and 100 to maximum discomfort.
Time Frame: baseline and 1 month [day 29]
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | CyclASol Ophthalmic Solution | Vehicle Ophthalmic Solution
Number analyzed (Participants) | 409 | 395
score on a scale | -12.2 (1.29) | -13.6 (1.31)

3. Secondary Outcome: Change From Baseline in Total Conjunctival Lissamine Green Staining
Description: Conjunctival staining was assessed by the investigator in the nasal and temporal sections. The Oxford Scheme was used for each section, with a possible score of 0-5 for each section, where 0=absent and 5=severe. The nasal and temporal scores were summed, for a possible score of 0-10 for each eye.
Time Frame: baseline and 1 month [day 29]
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | CyclASol Ophthalmic Solution | Vehicle Ophthalmic Solution
Number analyzed (Participants) | 409 | 395
score on a scale | -1.24 (0.078) | -0.91 (0.079)

4. Secondary Outcome: Proportion of Responders in Central Corneal Fluorescein Staining Score
Description: ≥ 1 score improvement for cCFS on National Eye Institute (NEI) scale: Central Corneal Fluorescein Staining (cCFS) is graded based on the NEI scale. The NEI scale divides the cornea in 5 subregions: central, inferior, superior, nasal, temporal. The score for each region ranges from 0-3; 0 corresponds to no staining (best), 3 corresponds to maximum staining (worst).
Time Frame: baseline and 1 month [day 29]
Measure: Count of Participants; unit: Participants
Arm/Group | CyclASol Ophthalmic Solution | Vehicle Ophthalmic Solution
Number analyzed (Participants) | 409 | 395
Participants | 275 | 238

5. Secondary Outcome: Proportion of Responders in Total Corneal Fluorescein Staining Score
Description: ≥ 3 scores improvement for tCFS on National Eye Insititute (NEI) scale: Total Corneal Fluorescein Staining (tCFS) is graded based on the NEI scale. The NEI scale divides the cornea in 5 subregions: central, inferior, superior, nasal, temporal. The score for each region ranges from 0-3; 0 corresponds to no staining (best), 3 corresponds to maximum staining (worst). The total score is the sum of the 5 subregions ranging from 0 (best) -15 (worst).
Time Frame: baseline and 1 month [day 29]
Measure: Count of Participants; unit: Participants
Arm/Group | CyclASol Ophthalmic Solution | Vehicle Ophthalmic Solution
Number analyzed (Participants) | 409 | 395
Participants | 293 | 236

6. Secondary Outcome: Change From Baseline in Central Corneal Fluorescein Staining
Description: Central Corneal Fluorescein Staining (cCFS) is graded based on the National Eye Institute (NEI) scale. The NEI scale divides the cornea in 5 subregions: central, inferior, superior, nasal, temporal. The score for each region ranges from 0-3; 0 corresponds to no staining (best), 3 corresponds to maximum staining (worst).
Time Frame: baseline and 1 month [day 29]
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | CyclASol Ophthalmic Solution | Vehicle Ophthalmic Solution
Number analyzed (Participants) | 409 | 395
score on a scale | -0.79 (0.045) | -0.67 (0.046)

7. Secondary Outcome: Change From Baseline in Total Corneal Fluorescein Staining
Description: as for outcome 1
Time Frame: baseline and 2 weeks [day 15]
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | CyclASol Ophthalmic Solution | Vehicle Ophthalmic Solution
Number analyzed (Participants) | 418 | 403
score on a scale | -3.53 (0.144) | -2.97 (0.147)

8. Secondary Outcome: Change From Baseline in Visual Analogue Scale (VAS) for Blurred Vision
Description: Blurred vision score is rated on a visual analogue scale (VAS) ranging from 0-100; 0 corresponds to no discomfort and 100 to maximum discomfort.
Time Frame: baseline and 1 month [day 29]
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | CyclASol Ophthalmic Solution | Vehicle Ophthalmic Solution
Number analyzed (Participants) | 409 | 395
score on a scale | -7.1 (1.19) | -6.1 (1.21)

ADVERSE EVENTS:
Time Frame: Adverse event data was were collected over the study period (29 days)
Arm/Group | CyclASol Ophthalmic Solution | Vehicle Ophthalmic Solution
All-Cause Mortality (participants affected / at risk) | 0/423 | 0/411
Serious Adverse Events (participants affected / at risk) | 2/423 | 3/411
Other Adverse Events (participants affected / at risk) | 45/423 | 37/411
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CyclASol Ophthalmic Solution (N=423) | Vehicle Ophthalmic Solution (N=411)
Partial Bowel Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Herpes Simplex Virus (Infections and infestations) | 0 (0) | 1 (1)
Left Foot Infection (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CyclASol Ophthalmic Solution (N=423) | Vehicle Ophthalmic Solution (N=411)
Instillation Site Pain (General disorders) | 45 | 37 — Administration site conditions

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-15): https://cdn.clinicaltrials.gov/large-docs/29/NCT04523129/Prot_SAP_000.pdf